CLINICAL TRIAL: NCT01030835
Title: Screening Protocol for the Evaluation of Research Participants at MPRC
Brief Title: Screening Protocol for the Evaluation of Research Participants at the Maryland Psychiatric Research Center (MPRC)
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909444; 09-DA-N444
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-10

CONDITIONS: Substance Use Disorders
Keywords: Screening Protocol; Comorbidity; Normal Controls; Substance Use Disorders; Substance Abuse Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- The National Institute of Drug Abuse (NIDA) is interested in developing a pool of potential research participants who may be eligible for research studies on drug abuse and addiction, pharmacological and psychosocial therapies for substance addiction, drug abuse and co-occurring psychiatric disorders, and the long-term effects of drugs on the development, function, and structure of the brain and other organ systems. To develop this pool of potential participants, researchers intend to screen individuals who may be eligible for future research studies.

Objectives:

- To identify, recruit, and screen participants for NIDA collaborative research protocols.

Eligibility:

- Individuals 18 years of age and older who are able to provide informed consent.

Design:

* Eligible participants will undergo two screening interviews: a telephone interview and an in-person interview. The phone interview will determine eligibility for the in-person interview.
* The in-person interview, which may require up to five visits to the clinical center, will involve any or all of the following procedures: (1) full physical examination and medical history; (2) psychiatric interview; (3) psychological testing; (4) electrocardiogram; (5) samples of blood, urine, and hair; and (6) other minimally invasive procedures as directed by the research staff.
* Participants will provide a photograph for confirmation of identity for subsequent visits and protocols.
* No clinical care will be provided under this protocol.

DETAILED DESCRIPTION:
The MPRC/NIDA collaborative research program attempts to: elucidate the nature of serious mental illnesses, drug abuse and addiction; determine the potential use of new therapies, both pharmacological and psychosocial; and decipher the long-term effects of drugs of abuse on the development, maturation, function, and structure of the brain and other organ systems. In support of this work, the scientific goal of this screening protocol is to assess potential research participants' eligibility for research studies. Screening will include medical and psychological tests and procedures. The data collected during screening are a unique and valuable source of information that aids in the research mission. Therefore, a secondary goal of this protocol is to obtain data that characterizes the population of subjects contacting NIDA about research participation and to analyze data so obtained, such as that on the prevalence and consequences of HIV/AIDS, viral hepatitis, and related diseases and issues of selection and sample bias in clinical research.

The screening process will be done in two stages, a telephone interview and an in-person evaluation. The telephone interview will last approximately 20 minutes and be conducted solely via the NIDA call center. Answers provided during the phone interview will indicate whether a caller is eligible for in-person screening. Those who appear eligible will be given an appointment at either NIDA or MPRC. This protocol pertains only to the in-person participants at MPRC. Written informed consent will be obtained when the person arrives. The screening process can involve up to 5 visits to MPRC.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults (at least age 18)
  2. Ability to understand and answer the questions posed

EXCLUSION CRITERIA:

1. Inability to provide valid informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2009-05-28; Study Completion 2012-04-10

CONTACTS AND LOCATIONS:
Overall Officials: David A Gorelick, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland
  - Maryland Psychiatric Research Center (MPRC) 55 Wade Avenue, Catonsville, Maryland